CLINICAL TRIAL: NCT05890443
Title: Mobile Application-Based Exercise Program Effects on Quality Of Life ın COPD; Randomized Experimental Study
Brief Title: Mobile-Application Based Respiratory Rehabilitation For COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Collaborators: Inonu University (Other)
Responsible Party: Principal Investigator, Ayten, Phd,Rn,lecturer, Ordu University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Project ID-TDK-2020-2048; Project ID-TDK-2020-2048 (Other Grant/Funding Number: İnonu unıversıty)
Record Dates: First submitted 2023-05-08; First posted 2023-06-06 (Actual); Last update posted 2023-06-06 (Actual); Status verified 2023-05

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Health-Related Quality Of Life; Dyspnea
Keywords: Dyspnea; Mobile Application; Quality Of Life,; Tele-rehabilitation; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Dyspnea | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: A Randomized Experimental Study
Who Masked: Participant
Masking Description: Experimental and control groups were evaluated separately. There was no need for blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group exercised via mobile application (Experimental): Individuals aged 40 and over with COPD were included in the study, while individuals with communication, mental, neurological and cognitive problems and unable to exercise were excluded from the study. Among those who met the inclusion criteria, those who had a smart-phone were assigned to the experimental group.
  Interventions: Behavioral: Exercise
- The group not included in the exercises via the mobile application. (No Intervention): Individuals aged 40 and over with COPD were included in the study. The individuals with communication, mental, neurological and cognitive problems and unable to exercise were excluded from the study. Those who did not have a smart-phone were assigned to the control group.

INTERVENTIONS:
Behavioral: Exercise — Before starting the research, self-management training in rehabilitation was given to both groups. While the exercise practices were carried out in the experimental group, encouraging reminders were made by following the background web page created in the experimental group.
  Other Names: self-management training
  Arms: Group exercised via mobile application

SUMMARY:
Abstract Purpose: This study aimed to determine the effect of mobile application-based exercise programs on the quality of life and dyspnea of patients with chronic obstructive pulmonary disease. This study was designed experimentally with a randomized control group.

Methods: A total of 76 COPD patients were included in the study. Individuals aged 40 and over with COPD were included in the study, while individuals with communication, mental, neurological and cognitive problems and unable to exercise were excluded from the study. Among those who met the inclusion criteria, those who had a smart-phone were assigned to the experimental group, while those who did not have a smart-phone were assigned to the control group. Self-management training was given to all individuals in both the control and experimental groups. After the training, the Saint George Respiratory Questionnaire (SGRQ) and dyspnea tests were administered to both groups. After the rehabilitation exercise program developed for the patients in the experimental group was applied, the tests were repeated for all groups.

Results: The mean age of the patients in the study was 65.5708± 9 in the control group, while the mean age of the experimental group was 67.61± 9.93. While the Borg dyspnea scale results of the experimental group were 6.45± 1.90 in the first test, the post-test measurements were 5.16± 1.65 (t = 7.66, p = 0.00). SGRQ pre-test and post-test total scores were 50.78± 16.39 and 41.99±15.04, respectively, in the experimental group (t=6.80 and p=0.08).

Conclusion: Respiratory and muscle strengthening exercises applied with the support of the mobile application, positively affected the quality of life of patients with COPD.

DETAILED DESCRIPTION:
Mobile Application-Based Exercise Program Effects on Quality Of Life ın COPD; Randomized Experimental Study

1. Introduction Chronic Obstructive Pulmonary Disease (COPD), is a common progressive but treatable disease characterized by airway obstruction. Symptoms such as shortness of breath and fatigue, especially during exercise, lead to a decrease in physical activity and fitness of these patients. 1, 2 This decrease in activity causes deterioration in the health-related quality of life of the individual. The primary goal of effective COPD treatment is to reduce the patient's symptoms and future risks. Respiratory rehabilitation, a non-pharmacological treatment method, is a first-line management strategy in patients with COPD. These rehabilitation programs reduces shortness of breath, increases exercise capacity and improves health-related quality of life.3 However, limited number of patients can benefit from respiratory rehabilitation due to various reasons such as lack of resources and motivation as well as accessibility problems. The insufficient number of rehabilitation centers and the fact that most centers are located in city centers create a significant limitation. In this respect, telemedicine-based rehabilitation can significantly facilitate the access of elderly population who have difficulty leaving their homes and who do not have access to these services due to the aforementioned factors. 3, 4, 5 The studies in literature report that rehabilitation utilizing technology performed in the home environment significantly improves the exercise capacity and quality of life of patients. 6, 7, 8 In this study, the investigators aimed to develop an alternative rehabilitation program for patients with COPD who can't access traditional rehabilitation applications. The effects of this developed mobile application-based program on the participants were evaluated statistically.
2. Methods In the present study, a mobile application that provided breathing and strengthening exercise training was developed to support the self-management of populations with COPD and to ensure their participation and continuity in an exercise program in their home environment. This application was developed with an aim to improve the dyspnea levels of populations with COPD, increase their exercise capacity, and improve their quality of life.

The study was a pre-test-post-test experimental study. The study was conducted on populations with COPD who presented to the pulmonary diseases clinic in a state hospital in a province. The study was carried out between October 2019 and June 2021, and the patients were followed at home for 10 weeks after exercise and self-management training.

The population of the study consisted of participants who were diagnosed with COPD and had no physical disability for exercise. Power analysis was performed to calculate the sample size. When α error was considered as 0.05 and the effect size was considered as 0.8, the sample size was determined to be 68 patients with COPD (34 in the experimental and 34 in the control group) with 90% power. However, considering that there would be dropouts, forty participants were included in both of the groups.

Patient Involvement: Patients aged 40 and over with COPD, who did not participate in the PR program during the last year and volunteered to participate in the study were included in the study. Patients with communication, mental, neurological and cognitive problems and those with disabilities to exercise were excluded from the study. The group that had a smartphone, met the inclusion criteria and volunteered to participate in the study was assigned to the experimental group. Participants who did not have a smartphone but, met the inclusion criteria were assigned to the control group. In addition, randomization was not performed. Assignment procedures to control and experimental groups were made by the researchers.The participants , who applied to the clinic during the study and met the criteria were assigned to the experimental and control groups until the number was completed.

2.1. Outline of the Developed Mobile Application The application ran on Android operating systems. The information of the participants using the application was recorded in the Sql Server 2019 database running on a Windows Server. Training regarding arm and leg exercises as well as breathing exercises based on the Hairmyres Home Exercise program and home exercises recommended for patients with COPD on the website of the Thoracic Society 9 was included in the mobile application. Video recordings of the exercises were made using live mannequins and added to the system. Written explanations of the exercise were added below the videos. While collecting the study data, the APK (Android Package Kit, Google and Open Hand send Alliance, ABD) was installed on the phones of the individuals. The patients registered on the web page created in the backend, created user names and passwords, and were logged into the system. The exercise flow chart and durations developed for the application are shown in figure 1.

2.2. Data Collection In the experimental group, the dyspnea scale (Borg Dyspnea Scale), Modified Medical Research Counsel (mMRC) Dyspnea scales, sitting-rising test and Saint George Respiratory Questionnaire (SGRQ) were initially administered. The results obtained were recorded in the first evaluation part of the personal information form.

Modified Borg Dyspnea Scale This scale was developed to measure the effort spent during physical exercise. It consists of ten items describing the severity of dyspnea according to their. 10 mMRC Dyspnea Scale This scale is used for grading the effects of shortness of breath in daily activities. The mMRC is a five-item scale that assesses patients based on various movements that cause shortness of breath. 11 Sitting-rising Test This test is an objective performance evaluation test that can be performed using simple equipment such as a chair and stopwatch. 12

SGRQ This questionnaire consists of three sections: symptom, activity, and effects of the disease. The symptom section includes dyspnea, cough, sputum, and respiratory problems. The activity section investigates physical activities that are restricted due to shortness of breath. In the impact section, the effects of the disease on the daily life of the individual are assessed. The score range of the questionnaire is between 0 (perfect health) and 100 (most severe disease). A change of four units in the score is considered clinically significant. The total score is determined by adding up the scores of the three sections and dividing it by 100.

Before starting the exercise training, the patients were given a training presentation on self-management. These trainings were carried out face-to-face and together with the patient's relatives. The content of self-management training consisted of drug use, disease control, and the importance of exercise. After the training, the exercises included in the application were taught to the participants in the experimental group. After these trainings, the mobile application was installed on the smart phones of the experimental group. The participants performed extremity muscle strengthening exercises for 15 minutes on three separate days a week for 10 weeks and performed breathing exercises for 10 minutes on the other three separate days of the week. During this period, patients' compliance with the program was recorded on the web page created in the backend. Participants compliance were encouraged with the program by visiting them at home once a week or calling them by phone.

The control group was not provided with any training other than self-management training. Pre-test data were obtained using the Borg Dyspnea Scale, SGRQ, sitting-rising test and mMRC Dyspnea Scale measurements.

After 10 weeks, post-test data were obtained from the control and experimental groups using Borg Dyspnea Scale, SGRQ, sitting-rising test and mMRC Dyspnea Scale. The results were recorded in the second evaluation part of the personal information form. The flowchart of the research is shown in Figure 2.

2.3. Evaluation of Data The data obtained in the research were analyzed using Statistical Package for Social Sciences for Windows 25.0. Descriptive statistical methods (number, percentage, mean, and standard deviation) were used while evaluating the data. Conformity of data to normal distribution was tested with normality tests and kurtosis-skewness values. It was determined that the data showed normal distribution. Therefore, parametric tests were preferred. Independent samples t-test was used to compare quantitative variables between two independent groups, and dependent samples t-test was used to compare variables between dependent samples.

2. Results At the beginning of the study, new participants were recruited instead of those who wanted to leave the study. The main aim, was to carry out the study with 40 participants. However, in the later stages of the study, two people from each group were lost despite all the precautions. These losses, occurred due to not being able to connect and wanting to leave the study.

ELIGIBILITY:
Inclusion Criteria:

Participants;

* Beıng 40 years or older,
* Not to have partıcıpated ın the PR program durıng the last year,
* Volunteering to partıcıpate ın the study,
* Beıng dıagnosed wıth COPD,
* Not having a condition that prevents you from exercising,
* In addıtıon, for the experiment group, ıt ıs necessary to have a smart phone for hımself or a close person.

Exclusion Criteria:

* Participants; Have a communication problem,
* Having mental or neurological problems,
* Having arthritis, advanced cardiovascular disease, and critical pulmonary hypertension.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2021-06-15 (Actual)

PRIMARY OUTCOMES:
Dyspnea | 10 weeks
  Modified Medical Research Counsel (mMRC) and modified borg dyspnea scales were used to determine the effect of respiratory strengthening exercises.
  Modified borg dyspnea scale;This scale is used to measure the degree of difficulty in breathing. Individuals are asked to rate their shortness of breath between 0 and 10. 0 means that breathing does not cause any difficulty, and 10 points mean that shortness of breath is maximum.
  The mMRC (Modified Medical Research Council) Dyspnoea Scale is used to assess the degree of baseline functional disability due to dyspnoea.
  mMrc scale in daily activities a short scale used to rate the effects of shortness of breath.There is a scoring table between 0 and 4 points. 0 represents shortness of breath only during exercise, while 4 points; indicates the most severe shortness of breath.
Respiratory quality of life | 10 weeks
  St. George's Respiratory Questionnaire (SGRQ);Disease-specific instrument designed to measure impact on overall health, daily life, and perceived well-being in patients with obstructive airways disease.SGRQ This questionnaire consists of three sections: symptom, activity, and effects of the disease. The symptom section includes dyspnea, cough, sputum, and respiratory problems. The activity section investigates physical activities that are restricted due to shortness of breath. In the impact section, the effects of the disease on the daily life of the individual are assessed. The score range of the questionnaire is between 0 (perfect health) and 100 (most severe disease). A change of four units in the score is considered clinically significant. The total score is determined by adding up the scores of the three sections and dividing it by 100.

CONTACTS AND LOCATIONS:
Overall Officials: Seyhan ÇITLIK SARITAŞ, Study Director — undefined [undefined:seyhancitlik@hotmail.com]
Locations (2):
- Turkey (Türkiye) (2):
  - Ayten, Ordu, Altınordu
  - Seyhan Çıtlık SARITAŞ, Malatya, Battalgazi̇

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tsakanikas VD, Gatsios D, Dimopoulos D, Pardalis A, Pavlou M, Liston MB, Fotiadis DI. Evaluating the Performance of Balance Physiotherapy Exercises Using a Sensory Platform: The Basis for a Persuasive Balance Rehabilitation Virtual Coaching System. Front Digit Health. 2020 Nov 27;2:545885. doi: 10.3389/fdgth.2020.545885. eCollection 2020. PMID 34713032
- [Background] Troosters T, Blondeel A, Janssens W, Demeyer H. The past, present and future of pulmonary rehabilitation. Respirology. 2019 Sep;24(9):830-837. doi: 10.1111/resp.13517. Epub 2019 Mar 13. PMID 30868699
- [Result] Kosteli MC, Heneghan NR, Roskell C, Williams SE, Adab P, Dickens AP, Enocson A, Fitzmaurice DA, Jolly K, Jordan R, Greenfield S, Cumming J. Barriers and enablers of physical activity engagement for patients with COPD in primary care. Int J Chron Obstruct Pulmon Dis. 2017 Mar 28;12:1019-1031. doi: 10.2147/COPD.S119806. eCollection 2017. PMID 28405162
- [Result] Zhang F, Zhong Y, Qin Z, Li X, Wang W. Effect of muscle training on dyspnea in patients with chronic obstructive pulmonary disease: A meta-analysis of randomized controlled trials. Medicine (Baltimore). 2021 Mar 5;100(9):e24930. doi: 10.1097/MD.0000000000024930. PMID 33655957
- [Result] Shen L, Zhang Y, Su Y, Weng D, Zhang F, Wu Q, Chen T, Li Q, Zhou Y, Hu Y, Jiang X, Jin X, Zhang A, Li H. New pulmonary rehabilitation exercise for pulmonary fibrosis to improve the pulmonary function and quality of life of patients with idiopathic pulmonary fibrosis: a randomized control trial. Ann Palliat Med. 2021 Jul;10(7):7289-7297. doi: 10.21037/apm-21-71. PMID 34353031
- [Result] Stamenova V, Liang K, Yang R, Engel K, van Lieshout F, Lalingo E, Cheung A, Erwood A, Radina M, Greenwald A, Agarwal P, Sidhu A, Bhatia RS, Shaw J, Shafai R, Bhattacharyya O. Technology-Enabled Self-Management of Chronic Obstructive Pulmonary Disease With or Without Asynchronous Remote Monitoring: Randomized Controlled Trial. J Med Internet Res. 2020 Jul 30;22(7):e18598. doi: 10.2196/18598. PMID 32729843
- [Result] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633
- [Result] Aboumatar H, Naqibuddin M, Chung S, Chaudhry H, Kim SW, Saunders J, Bone L, Gurses AP, Knowlton A, Pronovost P, Putcha N, Rand C, Roter D, Sylvester C, Thompson C, Wolff JL, Hibbard J, Wise RA. Effect of a Hospital-Initiated Program Combining Transitional Care and Long-term Self-management Support on Outcomes of Patients Hospitalized With Chronic Obstructive Pulmonary Disease: A Randomized Clinical Trial. JAMA. 2019 Oct 8;322(14):1371-1380. doi: 10.1001/jama.2019.11982. PMID 31593271
- See also: Vaidya T, Chambellan A, De Bisschop C. Sit-to-stand tests for COPD: a literature review. Respir Med, 2017;128: 70-77 — https://doi.org/10.1016/j.rmed.2017.05.003
- See also: Kendrick KR, Baxi SC, Smith RM. "Usefulness of the modified 0-10 Borg scale in assessing the degree of dyspnea in patients with COPD and asthma." J Emerg Nurs, 26.3 (2000): 216-222. — https://doi.org/10.1016/S0099-1767(00)90093-X
- See also: Mbada CE ,Olaoye MI ,Dada OO , et al. Comparative efficacy of clinic-based and tele-rehabilitation application of mckenzie therapy in chronic low-back pain. Telerehab.019; 11: 41-58 — https://doi.org/10.5195/ijt.2019.6260
- See also: Demir G, Akkoca O, Doğan R, Saryal S, Karabiyikoğlu G. The evaluation of dyspnea and quality of life in COPD. Tuberk Toraks. 2003; 51: 365-372 — https://europepmc.org/article/med/15143383